CLINICAL TRIAL: NCT04756414
Title: Clinical Effectiveness of Exposure Based Cognitive Behavioral Group Therapy for IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Perjohan Lindfors, Principal investigator, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBS-Sabb
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Cognitive Behavior Therapy, IBS, Group Therapy, Exposure,
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Patients recieve treatment from standard protocol at a gastroenterology unit. No specific adjustments is made for study purposes. Baseline data is collected before treatment and then again after treatment (POST).
  Interventions: Behavioral: Exposure based face-to-face Cognitive Behavior Group Therapy

INTERVENTIONS:
Behavioral: Exposure based face-to-face Cognitive Behavior Group Therapy — See under detailed description

SUMMARY:
The aim of the study is to evaluate the effects of a specific Cognitive Behavioral treatment protocol for patients with IBS used in routine care at a gastroenterology unit in Stockholm. The research question is whether the treatment has the same effects in routine care as it has had in efficacy studies.

The treatment is given by licenced psychologists (with CBT training) face-to-face in groups of 4-7 participants and lasts for ten sessions (ten weeks, normally).

DETAILED DESCRIPTION:
IBS is a debilitating condition that affects approximately one out of eleven persons world wide. It is often called a functional disorder, a term used to characterize painful conditions, whose biological mechanisms are not fully understood.

Diagnosis is made based on symptoms and exclusion of other conditions rather than specific tests or biological markers.

Treatment usually starts with diet counselling and a change of eating habits. If symptoms persist, a physician can prescribe medication of different types. But for some patients neither change of diet, nor medication is sufficient. Some of these patients may benefit from psychological treatment. There are a few different psychological treatments that have been proven efficacious in clinical trials. Most researched is Cognitive Behavior Therapy (CBT).

Our study is a clinical effectiveness trial without a control group. The data comes from a gastroenterology clinic in Stockholm and is collected as part of the work with continous improvement at the clinic.

Patients with diagnosed IBS are offered group treatment with a specific CBT protocol developed by our research group at Karolinska Institutet. The treatment comprises 6 different modules and stretches over ten sessions. The modules are: 1. Information regarding the treatment, IBS and mindfulness. 2 Hypervigilance and anxiety. 3. Behaviors and thoughts. 4. Behavior change part one - toilet habits including exposure to feared situations. 5. Behavior change part two - exposure to symptoms and avoidance/control behaviors. 6. Summary and relapse prevention.

Group sizes range from 4-7 patients and the treatment is given by licenced psychologists who are employed at the clinic.

ELIGIBILITY:
Inclusion Criteria:

- Diagnosed with IBS

Exclusion Criteria:

* Severe psychiatric condition (for example severe depression, self injuring, psychosis, PTSD)
* Unable or unwilling to participate in group therapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Symptom Rating Scale for IBS Gastrointestinal Symptom Rating Scale - IBS version | Baseline to 10 veeks
  Change in gastrointestinal symptoms measured with a self-rating scale from baseline to 10 weeks, and from baseline to 9 months for analysis of effect.The GSRS-IBS have 13 items about weekly gastrointestinal symptoms like bloating, hard stool, abdominal pain etc. It is a seven-point Likert scale from 1 (no discomfort at all) to 7 (very severe discomfort). The GSRS-IBS has excellent psychometric properties with internal consistency between α = .74 (for abdominal pain) to α = .85 (for satiety).

SECONDARY OUTCOMES:
Quality of Life in persons with Irritable Bowel Syndrome (QOL-IBS) | Baseline to 10 veeks
  QOL-IBS consists of 34 items scored between 1 and 6 and the total score is transformed to a 0-100 scale, where 0 represents minimum quality of life and 100 represents maximum quality of life. The IBS-QOL shows high internal consistency (Cronbach's a = .95) and test-retest reliability. r = .86
Visceral Sensitivity Index (VSI) | Baseline to 10 veeks
  VSI is a measure of gastro-intestinal anxiety (i.e., distress, avoidance, and safety behaviors in response to IBS-related stimuli). The VSI contains 15 items, which are scored between 1 and 6, rendering a total score between 0 (minimum GSA) and 75 (maximum GSA). The VSI has demonstrated high internal consistency (Cronbach's a = .90-.92) and has been shown to be associated with symptom severity and diagnostic status of IBS and also to be a mediator of the effect of exposure-based CBT on IBS symptoms.
The Montgomery-Åsberg Depression Rating Scale (MADRS-S) | Baseline to 10 veeks
  MADRS-S consists of 9 items that can be rated between 0 and 6, yielding a result between 0 and 54, where a higher number indicates more severe symptoms of depression. The scale was developed in 1993 and has been widely used. It has demonstrated good psychometric properties with an internal consistency between Cronbach's a = .84-.91

CONTACTS AND LOCATIONS:
Overall Officials: Perjohan Lindfors, PhD, MD, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallen H, Ljotsson B, Svanborg C, Rydh S, Falk L, Lindfors P. Exposure based cognitive behavioral group therapy for IBS at a gastroenterological clinic - a clinical effectiveness study. Scand J Gastroenterol. 2022 Aug;57(8):904-911. doi: 10.1080/00365521.2022.2047220. Epub 2022 Mar 9. PMID 35260030